CLINICAL TRIAL: NCT00478647
Title: A Multicenter Open-Label Study of Gene-Activated® Human Glucocerebrosidase (GA-GCB) Enzyme Replacement Therapy in Patients With Type 1 Gaucher Disease Previously Treated With Imiglucerase
Brief Title: Study of GA-GCB Enzyme Replacement Therapy in Type 1 Gaucher Disease Patients Previously Treated With Imiglucerase
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TKT034; 2006-006304-11 (EudraCT Number)
Record Dates: First submitted 2007-05-23; First posted 2007-05-25 (Estimated); Results first posted 2010-09-02 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Gaucher Disease
Keywords: Acid beta-glucocerebrosidase; human; glucocerebrosidase; Gaucher disease; Enzyme Replacement Therapy; D-glucosyl-N-acylsphingosine glucohydrolase; glucosylceramidase; gene activation; beta-glucocerebrosidase
MeSH Terms: conditions — Gaucher Disease | interventions — Glucosylceramidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GA-GCB (velaglucerase alfa) (Experimental): 15-60 U/kg, every other week via intravenous infusion
  Interventions: Biological: GA-GCB (velaglucerase alfa)

INTERVENTIONS:
Biological: GA-GCB (velaglucerase alfa) — 15-60 U/kg, every other week via intravenous infusion
  Other Names: gene-activated® human glucocerebrosidase; VPRIV®; GA-GCB

SUMMARY:
Gaucher disease is a rare lysosomal storage disorder caused by the deficiency of the enzyme glucocerebrosidase (GCB). Due to the deficiency of functional GCB, glucocerebroside accumulates within macrophages leading to cellular engorgement, organomegaly, and organ system dysfunction. The purpose of this study is to evaluate the safety and efficacy of every other week dosing of GA-GCB (velaglucerase alfa) in participants with type 1 Gaucher disease who were previously treated with imiglucerase.

DETAILED DESCRIPTION:
Type 1 Gaucher disease, the most common form, accounts for more than 90% of all cases and does not involve the CNS. Typical manifestations of type 1 Gaucher disease include hepatomegaly, splenomegaly, thrombocytopenia, bleeding tendencies, anemia, hypermetabolism, skeletal pathology, growth retardation, pulmonary disease, and decreased quality of life. Gene-Activated® human glucocerebrosidase (GA-GCB; velaglucerase alfa) is produced in a continuous human cell line using proprietary gene-activation technology and has an identical amino acid sequence to the naturally occurring human enzyme. GA-GCB contains terminal mannose residues that target the enzyme to the macrophages-the primary target cells in Gaucher disease. This study was designed to determine the safety of GA-GCB in men, women, and children with Type 1 Gaucher disease who were previously treated with imiglucerase. Each participant's duration of treatment will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

Includes:

* The participant has a documented diagnosis of type 1 Gaucher disease, as determined by deficient glucocerebrosidase (GCB) activity relative to normal as measured in leukocytes or by genotype analysis and the participant/legal guardian is willing and able to provide written informed consent prior to initiating any study-related procedures
* The participant has received consistent treatment with imiglucerase at a dose ≤ 60 U/kg and ≥ 15 U/kg every other week for a minimum of 30 consecutive months. Participants who are anti-imiglucerase antibody positive will be allowed to enter this study
* The participant is at least 2 years of age
* Female participants of child-bearing potential agree to use a medically acceptable method of contraception. Male participants must agree to use a medically acceptable method of birth control
* Participant must be sufficiently co-operative to participate in the study as judged by the Investigator.

Exclusion Criteria:

Includes:

* The participant has type 2 or 3 Gaucher disease or is suspected of having type 3 Gaucher disease
* The participant has received treatment with any investigational drug or device within the 30 days prior to study entry; such use during the study is not permitted
* Participant is HIV positive
* Participant is hepatitis B/C positive
* The participant presents with sustained iron, folic acid and/or vitamin B12 deficiency-related anemia during Screening
* The participant, participant's parent(s), or participant's legal guardian(s) is/are unable to understand the nature, scope, and possible consequences of the study
* The participant has a significant comorbidity that might affect study data or confound the study results
* The participant is unable to comply with the protocol or is otherwise unlikely to complete the study, as determined by the Investigator
* The participant has experienced an anaphylactic/anaphylactoid reaction during treatment with imiglucerase
* The participant has received miglustat during the 6 months prior to study enrollment
* The participant has an active, clinically significant spleen infarction
* The participant has active, progressive bone necrosis
* The participant is a pregnant and/or lactating female

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-07-25 (Actual); Primary Completion 2009-06-26 (Actual); Study Completion 2009-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (15):
- United States (11):
  - Regional Metabolic Center, Los Angeles, California
  - Children's Hospital Oakland, Oakland, California
  - Emory University, Decatur, Georgia
  - Feinberg School of Medicine, Chicago, Illinois
  - Children's of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital and Clinic, Kansas City, Missouri
  - NYU School of Medicine, New York, New York
  - Cincinatti Children's Hospital, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
  - Medical Genetics/Pediatrics, Salt Lake City, Utah
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Shaare Zedek Medical Center, Jerusalem, Israel
- Children's Memorial Health Institute, Warsaw, Poland
- Hospital Universitario Miguel Servet, Zaragoza, Spain
- The Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Result] Zimran A, Pastores GM, Tylki-Szymanska A, Hughes DA, Elstein D, Mardach R, Eng C, Smith L, Heisel-Kurth M, Charrow J, Harmatz P, Fernhoff P, Rhead W, Longo N, Giraldo P, Ruiz JA, Zahrieh D, Crombez E, Grabowski GA. Safety and efficacy of velaglucerase alfa in Gaucher disease type 1 patients previously treated with imiglucerase. Am J Hematol. 2013 Mar;88(3):172-8. doi: 10.1002/ajh.23383. Epub 2013 Jan 22. PMID 23339116

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled on 25 July 2007 and the last participant completed on 26 June 2009. Participants received the same dose of velaglucerase alfa (GA-GCB) as their previous dose of imiglucerase (range- </= 60 Unit per kilogram (U/kg) - >/=15 U/kg) every other week via intravenous infusion.
Pre-assignment Details: Participant at least 2 years old with documented diagnosis of type 1 Gaucher disease.Consistent treatment(every other week at a dose ≤/= 60 U/kg and ≥/= 15 U/kg) with imiglucerase for a minimum of 30 consecutive months;same dose during the 6 months prior to study enrollment.Minor dosing interval variance was allowed per standard clinical practice.
Period: Overall Study
Arm/Group | GA-GCB (Velaglucerase Alfa)
Started | 40
Completed | 38 (Intent-to-Treat (ITT)=participants who have received at least 1 full or partial dose of study drug.)
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | GA-GCB (Velaglucerase Alfa)
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 27
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (18.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22
  Spain | 1
  Poland | 5
  Israel | 9
  United Kingdom | 3
Baseline hemoglobin concentration [Median (Full Range); unit: gram per deciliter (g/dL)] | 13.775 [10.40 to 16.45]
Baseline liver volume [Median (Full Range); unit: Percent (%) body weight] | 1.90 [1.4 to 3.9]
Baseline platelet count [Median (Full Range); unit: 10^9 per liter (10^9/L)] | 162.00 [29.0 to 399.0]
Baseline spleen volume [Median (Full Range); unit: Percent (%) body weight] | 0.50 [0.2 to 3.2]

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline to Week 53 in Hemoglobin Concentration
Time Frame: Week 53
Population: ITT population.
Measure: Mean (90% Confidence Interval); unit: g/dL
Arm/Group | GA-GCB (Velaglucerase Alfa)
Number analyzed (Participants) | 40
g/dL | -0.101 [-0.272 to 0.070]

2. Secondary Outcome: Percent Change From Baseline to Week 53 in Platelet Count
Time Frame: Week 53
Population: ITT population.
Measure: Mean (90% Confidence Interval); unit: percent (%) change
Arm/Group | GA-GCB (Velaglucerase Alfa)
Number analyzed (Participants) | 40
percent (%) change | 7.04 [0.54 to 13.53]

3. Secondary Outcome: Percent Change From Baseline to Week 51 in Normalized Liver Volume
Description: Liver volume has been normalized for percentage (%) of body weight. Liver size relative to body weight= (Liver volume [cc]/Body weight [kg])*100
Time Frame: Week 51
Population: ITT population.
Measure: Mean (90% Confidence Interval); unit: Percent (%) change
Arm/Group | GA-GCB (Velaglucerase Alfa)
Number analyzed (Participants) | 40
Percent (%) change | -0.03 [-2.62 to 2.56]

4. Secondary Outcome: Percent Change From Baseline to Week 51 in Normalized Spleen Volume
Description: Spleen volume has been normalized for percentage (%) of body weight. Spleen size relative to body weight= (Spleen volume [cc]/Body weight [kg])*100
Time Frame: Week 51
Population: ITT population. Four splenectomized participants were excluded.
Measure: Mean (90% Confidence Interval); unit: Percent (%) change
Arm/Group | GA-GCB (Velaglucerase Alfa)
Number analyzed (Participants) | 36
Percent (%) change | -5.56 [-10.77 to -0.35]

5. Primary Outcome: Participants Who Experienced at Least One Adverse Event
Description: Safety was assessed throughout the study by assessments including adverse events, concomitant medication use, and vital signs. Additional safety assessments, including 12-lead ECGs, physical examinations, clinical laboratory tests and determination of the presence of anti-velaglucerase alfa antibodies. Refer to Adverse event section for further details.
Time Frame: Week 53
Population: Safety population included subjects who have received at least 1 full or partial dose of study drug.
Measure: Number; unit: participants
Arm/Group | GA-GCB (Velaglucerase Alfa)
Number analyzed (Participants) | 40
participants | 34

ADVERSE EVENTS:
Time Frame: Time of informed consent until 30 days after the last dose and/or until the event was resolved/stabilized or outcome was reached, whichever came first. Participants who discontinued/withdrew prior to Week 53, and followed up to 30 days after last dose.
Arm/Group | GA-GCB (Velaglucerase Alfa)
Serious Adverse Events (participants affected / at risk) | 4/40
Other Adverse Events (participants affected / at risk) | 31/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GA-GCB (Velaglucerase Alfa) (N=40)
Anaphylactoid reaction (Immune system disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GA-GCB (Velaglucerase Alfa) (N=40)
Hypertension (Vascular disorders) | 3 (15)
Fatigue (General disorders) | 5 (13)
Influenza like illness (General disorders) | 4 (5)
Malaise (General disorders) | 2 (33)
Non-Cardiac chest pain (General disorders) | 2 (3)
Pyrexia (General disorders) | 5 (7)
Anxiety (Psychiatric disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Blood glucose increased (Investigations) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 12 (29)
Paraesthesia (Nervous system disorders) | 3 (3)
Conjunctivitis (Eye disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 5 (11)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4)
Toothache (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (10)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (3)
Bronchitis (Infections and infestations) | 3 (4)
Influenza (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 8 (10)
Pharyngitis (Infections and infestations) | 2 (2)
Rhinovirus infection (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 5 (7)
Urinary tract infection (Infections and infestations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤180 days from the time submitted to Shire for review. Shire does not prohibit publication, but can require the removal of confidential information (excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication.